CLINICAL TRIAL: NCT06683599
Title: SEALion: a Study on the Effectiveness of Additional Oxygenation in Little Children During Intubation Using Oxygenation Delivered by Nasal Cannula
Brief Title: SEALion: Study on Supplemental Oxygenation Via Nasal Cannula for Young Children During Intubation
Acronym: SEALION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vinícius C Quintão, MD, MSc, PhD (Other)
Collaborators: University of Bern (Other); The University of Western Australia (Other)
Responsible Party: Sponsor-Investigator, Vinícius C Quintão, MD, MSc, PhD, Assistant Professor, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SEALION
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Difficult Airway; Difficult Airway Intubation; Neonate
Keywords: Difficult intubation; Apneic oxygenation; Neonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Tracheal intubation performed with a video laryngoscope with Miller-blade or Macintosh-blade size No. 0 or No. 1 without apneic oxygenation.
- Apneic oxygenation (Experimental): 1 L/kg/min FiO2 1.0 low-flow nasal supplemental oxygen with conventional nasal cannula during tracheal intubation performed with a video laryngoscope with Miller-blade or Macintosh-blade size No. 0 or No. 1.
  Interventions: Procedure: Apneic oxygenation

INTERVENTIONS:
Procedure: Apneic oxygenation — 1 L/kg/min FiO2 1.0 low-flow nasal supplemental oxygen with conventional nasal cannula during tracheal intubation performed with a video laryngoscope with Miller-blade or Macintosh-blade size No. 0 or No. 1.
  Arms: Apneic oxygenation

SUMMARY:
Tracheal intubation in neonates can be technically challenging, even for experienced pediatric anesthesiologists, with a high first-attempt success rate crucial to ensure safety. Intubation, while life-saving for children with circulatory shock or respiratory failure, carries risks of severe desaturation that can lead to hypoxic encephalopathy, cardiac arrest, or death. Neonates, especially, are prone to hypoxemia due to high oxygen consumption, low functional residual capacity, small closing capacity, and increased risk of airway collapse, which is exacerbated under anesthesia and neuromuscular paralysis. Rapid desaturation occurs after cessation of ventilation, with neonates facing shorter apnea times before desaturation. Studies show that about two-thirds of neonates undergoing non-emergency nasotracheal intubation experience desaturation (SpO₂ <80% for over 60 seconds), although low-flow oxygen supplementation (0.2 L/kg/min) can extend safe apnea time.

This study aims to investigate apneic oxygenation with VL (using Miller or Macintosh blades size 0 or 1) in operating rooms or intensive care units. We hypothesize that supplemental oxygen and standardized VL use will improve first-pass success rates and reduce adverse events.

DETAILED DESCRIPTION:
Eligible children will undergo preparation for intubation following the local Standard Operating Procedures (SOPs) of the pediatric anesthesia departments. Mandatory monitoring includes pulse oximetry (SpO2), heart rate (HR), and non-invasive blood pressure (NIBP).

Anesthesia Induction:

Where feasible, all children enrolled in this protocol will be pre-oxygenated for one minute prior to induction of anesthesia using a face mask with FiO2 1.0 and a flow rate of 6-10 L/min. Anesthesia induction for tracheal intubation will involve a combination of sedative or hypnotic drugs, opioids, and a non-depolarizing muscle relaxant.

Required Medications (per protocol):

Neuromuscular Blocking Agent (NMBA): One of the following-Rocuronium 0.5-1 mg/kg, Cis-Atracurium 0.2-0.5 mg/kg, Atracurium 0.5 mg/kg, Vecuronium 0.1 mg/kg, Mivacurium 0.2-0.3 mg/kg, or Succinylcholine 2 mg/kg.

Hypnotic Agent: One or more of the following-Thiopentone 4-7 mg/kg, Ketamine 0.5-2 mg/kg, Propofol 1-4 mg/kg, Midazolam 0.5-1 mg/kg, or Sevoflurane up to 8%.

Optional Medications: An opioid and/or anticholinergic may be administered at the anesthetist's discretion.

Pre-Intubation Preparation:

Following induction of anesthesia and administration of an NMBA, bag-mask ventilation with FiO2 1.0 (flow rate of 6-10 L/min) will be performed for 60 seconds until apnea occurs. To facilitate airway management, complete neuromuscular blockade will be confirmed using train-of-four (TOF) monitoring. Oxygen administration, laryngoscopy, and tracheal intubation will follow.

Intubation Procedure:

Oxygen administration during intubation is mandatory for all participants and will be randomized as follows:

Apneic Oxygenation: Oxygen will be administered at 1 L/kg/min via a conventional nasal cannula. Laryngoscopy and tracheal intubation will proceed following apneic oxygenation.

Standard Care: No apneic oxygenation will be administered. After induction, laryngoscopy and tracheal intubation will proceed without additional oxygen support.

Tube Selection:

For premature neonates under 1 kg, an uncuffed tube with an internal diameter (ID) of 2.5 will be used.

For premature neonates and newborns between 1 kg and 3.0 kg, an uncuffed tube with ID 3.0 will be used.

For babies over 3.0 kg up to 8 months, a cuffed tube with ID 3.0 or an uncuffed tube with ID 3.5 will be used.

For infants aged 8 to 12 months, a cuffed tube with ID 3.5 or an uncuffed tube with ID 4.0 will be used.

Oxygen delivery will follow the assigned randomization group, either via conventional nasal cannula (apneic oxygenation) or standard care.

Laryngoscope Blade Selection:

For children weighing less than 1 kg, a Miller or Macintosh blade, size No. 0, will be used. In cases of unexpected difficult intubation, the difficult airway algorithm will be applied. After an unsuccessful first intubation attempt with the assigned flow rate, clinical judgment will guide the intubating physician on whether to repeat the attempt with the same flow rate or to modify the flow rate, blade size, or type of laryngoscope. A maximum of four intubation attempts will be allowed, with the final attempt performed by the most experienced physician present. Additional tools, such as a stylet or bougie, may be used at any stage. If intubation remains unsuccessful, the difficult airway algorithm will be applied, and a supraglottic airway (SGA) device will be inserted.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients requiring oral or nasal tracheal intubation for elective, semi-elective, or urgent surgical and non-surgical procedures.
* Neonates and infants up to 52 weeks post-conceptual age.
* Written informed consent provided by legal guardians prior to the intervention.

Exclusion Criteria:

* Prediction of difficult intubation based on physical examination or a history of previous difficult intubation.
* Requirement for an alternative technique to direct laryngoscopy to secure the airway.
* Specific conditions, such as congenital heart disease requiring FiO₂ < 1.0, or cardiopulmonary collapse necessitating advanced life support and intubation for emergency surgical or non-surgical interventions.

Ages: 1 Minute to 52 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
First-attempt success rate | From randomization until up to 15 minutes
  The primary study outcome is to evaluate the first attempt success rate of oral tracheal intubation without desaturation (< 90%) and/or bradycardia (< 100 bpm) with video laryngoscope with supplemental oxygen (apneic oxygenation) vs without supplemental oxygen in infants up to 52 weeks postconceptual age. A successful tracheal intubation (ETI) attempt is defined as successful placement of a tracheal tube in the trachea, confirmed by visualization of the tube passing the vocal cords, a waveform capnography suggesting correct ETT placement and auscultation of breath sounds in the lungs

SECONDARY OUTCOMES:
Desaturation rate | From randomization until up to 15 minutes
  Occurrence and duration of moderate and severe desaturation (SpO2 < 90% and SpO2 < 80%), with or without bradycardia, during intubation.
Overall number of intubation attempts | From randomization until up to 15 minutes
  The overall number of intubation attempts.
Time to intubation | From randomization until up to 5 minutes
  Time required for intubation (in seconds, defined from the first introduction of laryngoscope between the lips till successful lung ventilation defined as positive capnography).
Respiratory complications rate | From randomization until up to 24 hours
  Respiratory complications and complications of airway management within the first 24 hours, such as airway injury, cardiopulmonary resuscitation, bleeding, aspiration of gastric contents, post-extubation stridor, laryngospasm, bronchospasm, need for High Flow Nasal Oxygen (if not preoperatively on oxygen), need for low flow nasal oxygen (if not preoperatively on oxygen) or need for re-intubation will be recorded. Respiratory complications are defined as the need for re-intubation after being extubated, persistent stridor (even if oxygen is not required), respiratory failure, the occurrence of pneumothorax, or the need for any additional diagnostic examination following respiratory problems (i.e., bronchoscopy, radiology).
First EtCO2 after successful intubation | From randomization until up to 10 minutes
  Value in mmHg or kPa of the first reliable etCO2 reading after successful intubation
Cormack-Lehane score | From randomization until up to 5 minutes
  The Cormack-Lehane score, classified as 1, 2a, 2b, 3, or 4, recorded at each laryngoscopy attempt
The need for additional devices | From randomization until up to 5 minutes
  The need for additional devices used at any step of intubation
Duration of severe desaturation | From randomization until up to 15 minutes
  Duration of moderate and severe desaturation (SpO2 < 80%), with or without bradycardia, during intubation
Percentage of Glottic Opening (POGO) score | From randomization until up to 5 minutes
  Percentage of Glottic Opening (POGO) score recorded at each laryngoscopy attempt, ranging from 0% to 100%, with 100% indicating the best possible glottic view

CONTACTS AND LOCATIONS:
Overall Officials: Vinicius C Quintao, MD, MSc, PhD, Principal Investigator — Hospital das Clinicas, Faculdade de Medicina, Universidade de Sao Paulo
Locations (3):
- Perth Children's Hospital, Perth, Western Australia, Australia
- Hospital das Clinicas HCFMUSP, São Paulo, Brazil
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durrmeyer X, Breinig S, Claris O, Tourneux P, Alexandre C, Saliba E, Beuchee A, Jung C, Levy C, Marchand-Martin L, Marcoux MO, Dechartres A, Danan C; PRETTINEO Research Group. Effect of Atropine With Propofol vs Atropine With Atracurium and Sufentanil on Oxygen Desaturation in Neonates Requiring Nonemergency Intubation: A Randomized Clinical Trial. JAMA. 2018 May 1;319(17):1790-1801. doi: 10.1001/jama.2018.3708. PMID 29715354
- [Background] Patel R, Lenczyk M, Hannallah RS, McGill WA. Age and the onset of desaturation in apnoeic children. Can J Anaesth. 1994 Sep;41(9):771-4. doi: 10.1007/BF03011582. PMID 7954992
- [Background] Hardman JG, Wills JS. The development of hypoxaemia during apnoea in children: a computational modelling investigation. Br J Anaesth. 2006 Oct;97(4):564-70. doi: 10.1093/bja/ael178. Epub 2006 Jul 27. PMID 16873387
- [Background] Schwartz DE, Matthay MA, Cohen NH. Death and other complications of emergency airway management in critically ill adults. A prospective investigation of 297 tracheal intubations. Anesthesiology. 1995 Feb;82(2):367-76. doi: 10.1097/00000542-199502000-00007. PMID 7856895
- [Background] Shiima Y, Berg RA, Bogner HR, Morales KH, Nadkarni VM, Nishisaki A; National Emergency Airway Registry for Children Investigators. Cardiac Arrests Associated With Tracheal Intubations in PICUs: A Multicenter Cohort Study. Crit Care Med. 2016 Sep;44(9):1675-82. doi: 10.1097/CCM.0000000000001741. PMID 27071070
- [Background] Stinson HR, Srinivasan V, Topjian AA, Sutton RM, Nadkarni VM, Berg RA, Raymond TT; American Heart Association Get With the Guidelines-Resuscitation Investigators. Failure of Invasive Airway Placement on the First Attempt Is Associated With Progression to Cardiac Arrest in Pediatric Acute Respiratory Compromise. Pediatr Crit Care Med. 2018 Jan;19(1):9-16. doi: 10.1097/PCC.0000000000001370. PMID 29135805
- [Background] Nishisaki A, Ferry S, Colborn S, DeFalco C, Dominguez T, Brown CA 3rd, Helfaer MA, Berg RA, Walls RM, Nadkarni VM; National Emergency Airway Registry (NEAR); National Emergency Airway Registry for kids (NEAR4KIDS) Investigators. Characterization of tracheal intubation process of care and safety outcomes in a tertiary pediatric intensive care unit. Pediatr Crit Care Med. 2012 Jan;13(1):e5-10. doi: 10.1097/PCC.0b013e3181fe472d. PMID 21057359
- [Background] Khemani RG, Markovitz BP, Curley MAQ. Characteristics of children intubated and mechanically ventilated in 16 PICUs. Chest. 2009 Sep;136(3):765-771. doi: 10.1378/chest.09-0207. Epub 2009 Jun 19. PMID 19542258
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Disma N, Virag K, Riva T, Kaufmann J, Engelhardt T, Habre W; NECTARINE Group of the European Society of Anaesthesiology Clinical Trial Network; AUSTRIA (Maria Vittinghoff); BELGIUM (Francis Veyckemans); CROATIA (Sandra Kralik); CZECH REPUBLIC (Jiri Zurek); DENMARK (Tom Hansen); ESTONIA (Reet Kikas); FINLAND (Tuula Manner); FRANCE (Christophe Dadure, Anne Lafargue); GERMANY (Karin Becke, Claudia Hoehne); GREECE (Anna Malisiova); HUNGARY (Andrea Szekely); IRELAND (Brendan O'Hare); ITALY (Nicola Disma); LATVIA (Zane Straume); LITHUANIA (Laura Lukosiene); LUXEMBOURG (Bernd Schmitz); MALTA (Francis Borg); NETHERLANDS (Jurgen de Graaff); NORWAY (Wenche B Boerke); POLAND (Marzena Zielinska); PORTUGAL (Maria Domingas Patuleia); ROMANIA (Radu Tabacaru); SERBIA (Dusica Simic); SLOVAKIA (Miloslav Hanula); SLOVENIA (Jelena Berger); SPAIN (Ignacio Galvez Escalera); SWEDEN (Albert Castellheim); SWITZERLAND (Walid Habre); TURKEY (Dilek Ozcengiz - Zehra Hatipoglu); UKRAINE (Dmytro Dmytriiev); UNITED KINGDOM (Thomas Engelhardt, Suellen Walker); Management Team. Difficult tracheal intubation in neonates and infants. NEonate and Children audiT of Anaesthesia pRactice IN Europe (NECTARINE): a prospective European multicentre observational study. Br J Anaesth. 2021 Jun;126(6):1173-1181. doi: 10.1016/j.bja.2021.02.021. Epub 2021 Apr 1. PMID 33812665
- [Background] Hodgson KA, Owen LS, Kamlin COF, Roberts CT, Newman SE, Francis KL, Donath SM, Davis PG, Manley BJ. Nasal High-Flow Therapy during Neonatal Endotracheal Intubation. N Engl J Med. 2022 Apr 28;386(17):1627-1637. doi: 10.1056/NEJMoa2116735. PMID 35476651